CLINICAL TRIAL: NCT04111432
Title: A Randomized, Controlled Clinical Trial to Evaluate the Safety and Immunogenicity of Concomitant Administration of EV71 Vaccine With Measles, Mumps, and Rubella Combined Live Attenuated Vaccine/ Encephalitis Live Attenuated Vaccine
Brief Title: Safety and Immunogenicity of Concomitant Administration of EV71 Vaccine With Expanded Programme on Immunization Vaccines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Collaborators: Shaanxi Provincial Center for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EV71-SN-2019-01
Record Dates: First submitted 2019-09-29; First posted 2019-10-01 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Hand, Foot and Mouth Disease
Keywords: Inactivated Enterovirus Type 71 (EV71) Vaccine; Concomitant vaccination; Safety; Immunogenicity; Infant
MeSH Terms: conditions — Hand, Foot and Mouth Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I-EV71 and EPI vaccines Concomitant administration (Experimental): EV71 Vaccine (intramuscular injection,0.5ml,first dose)/measles mumps, and rubella combined live attenuated vaccine (subcutaneous injection,0.5ml) on day 0 and EV71 Vaccine (intramuscular injection, 0.5ml,second dose)/ encephalitis live attenuated vaccine (subcutaneous injection, 0.5ml) on day 30
  Interventions: Biological: Concomitant administration of EV71vaccine with EPI vaccines
- Group II-EPI vaccine only Single injection of EPI vaccine: (Active Comparator): measles mumps, and rubella combined live attenuated vaccine (subcutaneous injection,0.5ml) on day 0 and encephalitis live attenuated vaccine (subcutaneous injection, 0.5ml) on day 30
  Interventions: Biological: Single injection of EPI vaccine
- Group III-EV71 vaccine only EV71 Vaccine only (Active Comparator): the first and second dose of EV71 Vaccine (intramuscular injection,0.5ml) on day 0 andday 30 respectively
  Interventions: Biological: EV71 Vaccine only

INTERVENTIONS:
Biological: Concomitant administration of EV71vaccine with EPI vaccines — The investigated EV17 vaccine was manufactured by Sinovac Biotech Co., Ltd.# the MMR vaccine was manufactured by Shanghai Institute of Biological Products Co.,Ltd.; the Live attenuated Japanese encephalitis vaccine was manufactured by Chengdu Institute of Biological Products Co.,Ltd.
  Arms: Group I-EV71 and EPI vaccines Concomitant administration
Biological: Single injection of EPI vaccine — The MMR vaccine was manufactured by Shanghai Institute of Biological Products Co.,Ltd.; the Live attenuated Japanese encephalitis vaccine was manufactured by Chengdu Institute of Biological Products Co.,Ltd.
  Arms: Group II-EPI vaccine only Single injection of EPI vaccine:
Biological: EV71 Vaccine only — The investigated EV17 vaccine was manufactured by Sinovac Biotech Co., Ltd.
  Arms: Group III-EV71 vaccine only EV71 Vaccine only

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of concomitant administration of EV71 vaccine with measles mumps, and rubella combined live attenuated vaccine/ encephalitis live attenuated vaccine.

DETAILED DESCRIPTION:
This study is an open-label, single-center, randomized, comparative phase IV clinical trial. The purpose of this study is to evaluate the safety andimmunogenicity of concomitant administration of EV71 vaccine manufactured by Sinovac (Beijing) Vaccine Technology Co., Ltd. with measles mumps, and rubella combined live attenuated vaccine/ encephalitis live attenuated vaccine. 360 healthy infants of 8 months old as participants are randomly assigned into three experimental groups in the ratio 1:1:1. The group I receive EV71 Vaccine (first dose)&measles mumps, and rubella combined live attenuated vaccine on day 0 and EV71 vaccine (second dose)&encephalitis live attenuated vaccine on day 30. The group II receive measles mumps, and rubella combined live attenuated vaccine on day 0 and encephalitis live attenuated vaccine on day 30. The group III receive the first and second dose of EV71 Vaccine on day 0 and day 30 respectively.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer aged ≥ 8 months;
* Proven legal identity;
* Guardians of the participants should be capable of understanding the written consent form, and such form should be signed before the infant being included into this study.

Exclusion Criteria:

* Prior vaccination with EV71 vaccine;
* Prior vaccination with MMR vaccine or vaccine including mumps or measles or mumps or rubella vaccine components;
* Prior vaccination with Encephalitis B vaccine；
* Cannot be vaccinated with both arms at the same time；
* History of hand，foot and mouth disease;
* History of measles or mumps or rubella or encephalitis B；
* Allergy to gentamicin; history of allergy to any vaccine or vaccine ingredient, or serious adverse reaction(s) to vaccination, such as urticaria,difficulty in breathing, angioneurotic edema, pain, etc;
* Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc;
* Autoimmune diseases or immunodeficiency/immunosuppression;
* Severe neurological disorders (epilepsy, convulsions or convulsions) or psychosis;
* History of thyroidectomy, absence of spleen, functional absence of spleen, and any circumstances leading to absence of spleen or splenectomy;
* Diagnosed coagulation function abnormal (e.g., coagulation factor deficiency, coagulation disorder, or platelet abnormalities) , or obvious bruising or coagulation disorders;
* Any immunosuppressant, cytotoxic medicine, or inhaled corticosteroids (except corticosteroid spray for treatment of allergic rhinitis or corticosteroid treatment on surface for acute non-complicated dermatitis) in the past 6 months;
* Receipt of any of the following products:

  1. Blood product within 3 months prior to study entry;
  2. Any live attenuated vaccine within 14 days prior to study entry;
  3. Any subunit vaccine or inactivated vaccine within 7 days prior to study entry;
  4. Any other study drugs within 30 days prior to study entry;
* Acute disease or acute stage of chronic disease within 7 days prior to study entry;
* Axillary temperature > 37.0#;
* Any other factor that suggesting the volunteer is unsuitable for this study based on the opinions of investigators.

Min Age: 8 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2019-07-26 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
The seroconversion rates（SCR） of the EV71 neutralizing antibody 30 days after two dose of EV71 vaccines | 30 days after two dose of EV71 vaccines
  Immunogenicity indicator

SECONDARY OUTCOMES:
The seroconversion rates（SCR） of the Measles IgG antibody，Rubella 30 IgG antibody and Mumps IgG antibody 60 days after one dose of MMR vaccine | 60 days after one dose of MMR vaccine
  Immunogenicity indicator
The seroconversion rates（SCR） of the Japanese encephalitis neutralizing antibody 30 days after one dose of Encephalitis B vaccine | 30 days after one dose of Encephalitis B vaccine
  Immunogenicity indicator
EV71 neutralizing antibody positive rate 30 days of two dose of EV71 vaccines | 30 days after two dose of EV71 vaccines
  Immunogenicity indicator
The Geometric mean titer (GMT) of the EV71 neutralizing antibody 30 days of two dose of EV71 vaccines | 30 days after two dose of EV71 vaccines
  Immunogenicity indicator
Measles IgG antibody，Rubella 30 IgG antibody and Mumps IgG antibody positive rate 60 days after one dose of MMR vaccine | 60 days after one dose of MMR vaccine
  Immunogenicity indicator
The Geometric mean titer (GMT) of Measles IgG antibody，Rubella 30 IgG antibody and Mumps IgG antibody 60 days after one dose of MMR vaccine | 60 days after one dose of MMR vaccine
  Immunogenicity indicator
The Japanese encephalitis neutralizing antibody positive rate 30 days after one dose of Encephalitis B vaccine | 30 days after one dose of Encephalitis B vaccine
  Immunogenicity indicator
The Geometric mean titer (GMT) of Japanese encephalitis neutralizing antibody 30 days after one dose of Encephalitis B vaccine | 30 days after one dose of Encephalitis B vaccine
  Immunogenicity indicator
Incidence of solicited local or systemic adverse events within 7 days or 14 days after each dose | 7 days or 14 days after each dose of injection
  Safety indicator
The incidences of adverse reactions after each does | 0-30 days after each dose
  After each dose, a 30-minute safety observation will be conducted immediately. The body temperature, solicited local and general adverse events (AE) on day 0-7 or day 0-14 were reported. Unsolicited adverse events on day 0-30 were also reported.
Incidence of serious adverse events (SAEs) during the period of safety monitoring | 0-30 days after each dose
  Serious adverse events (SAEs) will be collected during the period of safety monitoring after each dose

CONTACTS AND LOCATIONS:
Overall Officials: Shaobai Zhang, Principal Investigator — Shaanxi Provincal Center for Disease Control and Preventione
Locations (1):
- Hanbin District Center for Disease Control and Prevention, Ankang, Shaanxi, China